CLINICAL TRIAL: NCT04987892
Title: Investigating Medication vs. Prostatic Urethral Lift: Assessment and Comparison of Therapies for Benign Prostatic Hyperplasia
Brief Title: Investigating Medication vs. Prostatic Urethral Lift: Assessment and Comparison of Therapies for BPH
Acronym: IMPACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00014
Record Dates: First submitted 2021-07-09; First posted 2021-08-03 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: BPH
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prostatic Lift (Active Comparator): Treatment with the UroLift System
  Interventions: Device: UroLift System
- Medication (Active Comparator): Treatment with Tamsulosin HCl 0.4mg
  Interventions: Drug: Tamsulosin Hydrochloride

INTERVENTIONS:
Device: UroLift System — Prostatic lift
  Arms: Prostatic Lift
Drug: Tamsulosin Hydrochloride — Tamsulosin HCl 0.4mg
  Other Names: Flomax
  Arms: Medication

SUMMARY:
This prospective, multicenter, two-arm, 1:1 randomized controlled trial (RCT) will enroll approximately 250 males at approximately 25 sites located within the United States. All enrolled subjects will be 45 years of age or older diagnosed with symptomatic benign prostatic hyperplasia (BPH). They will be randomized to one of two readily available, marketed BPH therapies; Prostatic Urethral Lift procedure with the UroLift System (PUL Arm) or 0.4mg tamsulosin HCl (MED Arm).

DETAILED DESCRIPTION:
This prospective, multicenter, two-arm, 1:1 randomized controlled trial (RCT) will enroll approximately 250 males at approximately 25 sites located within the United States. All enrolled subjects will be 45 years of age or older diagnosed with symptomatic benign prostatic hyperplasia (BPH). They will be randomized to one of two readily available, marketed BPH therapies; Prostatic Urethral Lift procedure with the UroLift System (PUL Arm) or 0.4mg tamsulosin HCl (MED Arm).Men 45 or older diagnosed with symptomatic benign prostatic hyperplasia (BPH). BPH symptoms may range from mild (8) to severe (35) on the IPSS scale. All enrolled men must meet selection criteria and be candidates for therapy with both UroLift System and 0.4 mg tamsulosin HCl.

ELIGIBILITY:
Inclusion Criteria:

1. Male 45 years of age or older
2. Diagnosis of BPH
3. Experiencing symptoms of BPH as indicated by an IPSS ≥8 and ≤30
4. Willing to wash out of current BPH medication(s), as applicable
5. An appropriate candidate for both BPH therapies evaluated in this study.
6. Ability to understand and consent to participate in this study
7. Willing and able to participate in follow-up evaluations

Exclusion Criteria:

1. Use of alpha blocker for BPH unless washed-out for 30 days
2. Use of daily phosphodiesterase type 5 inhibitor (PDE5i) for BPH unless washed-out for 30 days
3. 5-alpha-reductase inhibitors for BPH used within 6 months of therapy initiation
4. Current urinary tract infection or prostatitis
5. Current gross hematuria
6. Urinary incontinence presumed due to incompetent sphincter
7. Catheter-dependent urinary retention within 1 month prior to enrollment
8. Prostate volume greater than 100 cc as measured by TRUS
9. Prostate specific antigen level of greater than 10 ng/ml within one year of enrollment unless prostate cancer has been ruled out
10. History of neurogenic or atonic bladder
11. History prostate cancer treatment
12. Known to be hypersensitive to tamsulosin HCl or any component of tamsulosin HCl capsules
13. Known allergy to nickel, titanium, or stainless steel
14. Prior minimally invasive or surgical intervention for BPH
15. Urethral conditions that may prevent insertion of delivery system into bladder.
16. Currently enrolled in any other investigational clinical research trial that has not completed the primary endpoint
17. History of medical, surgical or other conditions that, in the opinion of the investigator, would interfere with the treatment or evaluation of the subject

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be male. The study is evaluation the population of men diagnosed with benign prostatic hyperplasia.
Enrollment: 250 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Paired comparison of International Prostate Symptom Score (IPSS) percent change | 3 Months after Therapy Initiation
  The primary study analysis compares the change in BPH symptoms in the PUL Arm to the change in BPH symptoms in the MED Arm measured 3 months after BPH therapy initiation. This will be measure by International Prostate Symptom Score (IPSS) percent change. IPSS ranges from 0-35, healthier patients have lower scores than patients more effected by BPH symptoms.

SECONDARY OUTCOMES:
Change in Quality of Life (QoL) | 3 months after BPH Therapy Initiation
  The secondary analysis assesses the change in quality of life (QoL) due to urinary symptoms between the PUL and MED Arms measured 3 months after initiation of BPH therapy. This will be measured by change in QoL, ranging from 0-6. Healthier patients have lower scores than patients more effected by BPH symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roehrborn, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Neotract, Pleasanton, California, United States